CLINICAL TRIAL: NCT04649359
Title: MAGNETISMM-3 AN OPEN-LABEL, MULTICENTER, NON-RANDOMIZED PHASE 2 STUDY OF ELRANATAMAB (PF-06863135) MONOTHERAPY IN PARTICIPANTS WITH MULTIPLE MYELOMA WHO ARE REFRACTORY TO AT LEAST ONE PROTEASOME INHIBITOR, ONE IMMUNOMODULATORY DRUG AND ONE ANTI-CD38 ANTIBODY
Brief Title: MagnetisMM-3: Study Of Elranatamab (PF-06863135) Monotherapy in Participants With Multiple Myeloma Who Are Refractory to at Least One PI, One IMiD and One Anti-CD38 mAb
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1071003; MagnetisMM-3 (Other: Alias Study Number); 2023-504479-25-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2020-11-06; First posted 2020-12-02 (Actual); Results first posted 2023-10-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Multiple Myeloma; relapsed Multiple Myeloma; refractory Multiple Myeloma; PF-06863135; BCMA; bispecific; bispecific antibody; BCMA-CD3 bispecific; Elranatamab; MagnetisMM-3
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elranatamab (cohort A) (Experimental): BCMA-CD3 bispecific antibody
  Interventions: Drug: Elranatamab (PF-06863135)
- Elranatamab (cohort B) (Experimental): BCMA-CD3 bispecific antibody
  Interventions: Drug: Elranatamab (PF-06863135)

INTERVENTIONS:
Drug: Elranatamab (PF-06863135) — BCMA-CD3 bispecific antibody

SUMMARY:
The purpose of the study is to evaluate whether single-agent Elranatamab (PF-06863135) can provide clinical benefit in participants with relapsed/refractory multiple myeloma. Elranatamab is a bispecific antibody: binding of Elranatamab to CD3-expressing T-cells and BCMA-expressing multiple myeloma cells causes targeted T-cell-mediated cytotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma (IMWG criteria, Rajkumar et al, 2014)
* Measurable disease, as defined by at least 1 of the following:

  1. Serum M-protein >0.5 g/dL by SPEP
  2. Urinary M-protein excretion >200 mg/24 hours by UPEP
  3. Serum immunoglobulin FLC≥10 mg/dL (≥100 mg/L) AND abnormal serum immunoglobulin kappa to lambda FLC ratio
* Refractory to at least one IMiD
* Refractory to at least one PI
* Refractory to at least one anti-CD38 antibody
* Relapsed/refractory to last anti-myeloma regimen
* Cohort A: has not received prior BCMA-directed therapy
* Cohort B: has received prior BCMA-directed therapy (ADC or CAR T cells)
* ECOG performance status ≤2
* Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade ≤1
* Not pregnant and willing to use contraception

Exclusion Criteria:

* Smoldering multiple myeloma
* Active Plasma cell leukemia
* Amyloidosis
* POEMS syndrome
* Stem cell transplant within 12 weeks prior to enrollment
* Active HBV, HCV, SARS-CoV2, HIV, or any active, uncontrolled bacterial, fungal, or viral infection
* Any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ.
* Previous administration with an investigational drug within 30 days or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (86):
- United States (44):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - The Regents of the University of California, Irvine, California
  - Ronald Reagan UCLA Medical Center Drug information Center, Los Angeles, California
  - The Regents of the University of California, Los Angeles, California
  - UCLA Hematology/Oncology Clinic, Los Angeles, California
  - UCLA Ronald Reagan Medical Center, Los Angeles, California
  - UC Irvine Health - Chao Family Comprehensive Cancer Center, Orange, California
  - Baptist Hospital of Miami, Miami, Florida
  - Winship Cancer Institute @ Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northwestern Medical Group, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Loyola University Chicago performing research at Loyola University Medical Center, Maywood, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - State University of Iowa, Iowa City, Iowa
  - University of Iowa - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Cancer Institute, St. Matthews Campus, Louisville, Kentucky
  - Norton Women's and Children's Hospital, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hackensack University Medical Center, Edison, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Regional Cancer Care Associates, LLC, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center - Investigational Drug Service Pharmacy, Long Island City, New York
  - Memorial Sloan Kettering Cancer Center - David H. Koch Center for Cancer Care, New York, New York
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - Weill Cornell Medical College - New York-Presbyterian Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - St Francis Physician Services Inc, Greenville, South Carolina
  - St. Francis Hospital, Greenville, South Carolina
  - Saint Francis Hospital Cancer Center, Greenville, South Carolina
  - St Francis Eastside, Greenville, South Carolina
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Baylor University Medical Center, Baylor Scott & White, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
- Australia (4):
  - Epworth Healthcare, East Melbourne, Victoria
  - St Vincent's Hospital (Melbourne), Fitzroy, Victoria
  - The Alfred, Melbourne, Victoria
  - Epworth Healthcare, Richmond, Victoria
- Belgium (4):
  - ZNA-Middelheim, Antwerp
  - ZNA Stuivenberg, Antwerp
  - Universitair Ziekenhuis Antwerpen, Edegem
  - CHU UCL Namur site Godinne, Yvoir
- Canada (6):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Alberta Health Services and The Governors of The University of Alberta, Edmonton, Alberta
  - CIUSSS-EMTL, Installation Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre - Glen Site, Montreal, Quebec
- France (6):
  - CHU de Lille - Hopital Claude Huriez, Lille
  - CHU de Nantes - Hôtel Dieu, Nantes
  - Hopital Saint-Louis, Paris
  - Hôpital Saint-Antoine, Paris
  - Centre Hospitalier Lyon Sud - Service d'Hematologie Clinique, Pierre-Bénite
  - CHU de Poitiers, Pôle Régional de Cancérologie, Poitiers
- Germany (4):
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitätsklinikum Hamburg - Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinik Schleswig-Holstein, Kiel
- Japan (7):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Gunma University Hospital, Maebashi, Gunma
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Iwate Medical University Hospital, Yahaba-cho, Iwate
  - Tohoku University Hospital, Sendai, Miyagi
  - Japanese Red Cross Medical Center, Shibuya-ku, Tokyo
  - Yamagata University Hospital, Yamagata
- Poland (3):
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Szpital Uniwersytecki nr 2 im. dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Szpital Kliniczny im. Heliodora Święcickiego UM w Poznaniu, Poznan
- Spain (7):
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruna
  - Institut Catala d' Oncologia. Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Clinic de Barcelona, Barcelona
  - Clinica Universitaria de Navarra, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Doctor Peset, Valencia
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Elmeliegy M, Soltantabar P, Hibma J, Ashman O, Wang D, Lon HK. Elranatamab Fixed Dosing: A Safe, Effective, and Convenient Dosing Approach. Target Oncol. 2025 Sep;20(5):821-831. doi: 10.1007/s11523-025-01170-4. Epub 2025 Aug 19. PMID 40830740
- [Derived] Lon HK, Hibma J, Jiang S, Sullivan S, Vandendries E, Skoura A, Wang D, Elmeliegy M. Population Exposure-Response Efficacy Analysis of Elranatamab (PF-06863135) in Patients with Multiple Myeloma. Target Oncol. 2025 Sep;20(5):803-819. doi: 10.1007/s11523-025-01168-y. Epub 2025 Aug 18. PMID 40826257
- [Derived] Gordan LN, Bensimon AG, Mu F, Kim N, Wu B, Lin D, Paner A, Fowler J, Marshall A, Van Sanden S, Ammann E, Goble J, Zhang X, Le HH, Min EE, Garrison LP Jr. Cost per responder for teclistamab and elranatamab in relapsed or refractory multiple myeloma in the United States. J Med Econ. 2025 Dec;28(1):910-920. doi: 10.1080/13696998.2025.2514909. Epub 2025 Jun 14. PMID 40495704
- [Derived] Elmeliegy M, Viqueira A, Vandendries E, Hickman A, Conte U, Irby D, Hibma J, Lon HK, Piscitelli J, Soltantabar P, Skoura A, Jiang S, Wang D. Dose Optimization of Elranatamab to Mitigate the Risk of Cytokine Release Syndrome in Patients with Multiple Myeloma. Target Oncol. 2025 Mar;20(2):349-359. doi: 10.1007/s11523-025-01134-8. Epub 2025 Feb 25. PMID 40000533
- [Derived] Iida S, Ito S, Yokoyama H, Ishida T, Nagai Y, Handa H, Ito S, Kamei Y, Nakamura M, Suzuki K. Elranatamab in Japanese patients with relapsed/refractory multiple myeloma: results from MagnetisMM-2 and MagnetisMM-3. Jpn J Clin Oncol. 2024 Sep 4;54(9):991-1000. doi: 10.1093/jjco/hyae068. PMID 38794892
- [Derived] Mol I, Hu Y, LeBlanc TW, Cappelleri JC, Chu H, Nador G, Aydin D, Schepart A, Hlavacek P. A matching-adjusted indirect comparison of the efficacy of elranatamab versus physician's choice of treatment in patients with triple-class exposed/refractory multiple myeloma. Curr Med Res Opin. 2024 Feb;40(2):199-207. doi: 10.1080/03007995.2023.2277850. Epub 2024 Jan 24. PMID 38078866
- [Derived] Lesokhin AM, Tomasson MH, Arnulf B, Bahlis NJ, Miles Prince H, Niesvizky R, Rodriotaguez-Otero P, Martinez-Lopez J, Koehne G, Touzeau C, Jethava Y, Quach H, Depaus J, Yokoyama H, Gabayan AE, Stevens DA, Nooka AK, Manier S, Raje N, Iida S, Raab MS, Searle E, Leip E, Sullivan ST, Conte U, Elmeliegy M, Czibere A, Viqueira A, Mohty M. Elranatamab in relapsed or refractory multiple myeloma: phase 2 MagnetisMM-3 trial results. Nat Med. 2023 Sep;29(9):2259-2267. doi: 10.1038/s41591-023-02528-9. Epub 2023 Aug 15. PMID 37582952
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with relapsed/refractory multiple myeloma (RRMM), who were refractory to at least 1 proteasome inhibitor, 1 immunomodulatory drug, and 1 anti-cluster of differentiation38 (CD38) monoclonal antibody were included. Study enrolled participants into 2 independent and parallel cohorts: cohort A and B.
Pre-assignment Details: A total of 187 participants were enrolled and assigned to study treatment. Results are reported at primary completion date. Data for only those primary and secondary outcome measures whose analysis is complete and final have been reported. Data for remaining secondary outcome measures will be posted upon completion of analysis at secondary completion date.
Groups:
- Cohort A: Participants who had not previously received a B-cell maturation antigen (BCMA)-directed therapy (BCMA-naïve participants) received subcutaneous elranatamab with a priming regimen of 12 milligrams (mg) on Cycle 1 Day 1 and 32 mg on Cycle 1 Day 4 followed by 76 mg weekly thereafter starting from Cycle 1 Day 8. Each cycle was 28 days. Treatment was continued until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or study termination. If a participant had received weekly dosing (QW) for at least 6 cycles and had achieved a partial response (PR) or better persisting for at least 2 months, the dose interval was changed to once every 2 weeks (Q2W). The initial 4 enrolled participants received subcutaneous elranatamab with a priming regimen of 44 mg on Cycle 1 Day 1 followed by 76 mg weekly thereafter starting from Cycle 1 Day 8.
- Cohort B: Participants who had previously received a BCMA-directed therapy (BCMA-exposed) received subcutaneous elranatamab with a priming regimen of 12 milligrams (mg) on Cycle 1 Day 1 and 32 mg on Cycle 1 Day 4 followed by 76 mg weekly thereafter starting from Cycle 1 Day 8. Each cycle was 28 days. Treatment was continued until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or study termination. If a participant had received weekly dosing (QW) for at least 6 cycles and had achieved a partial response (PR) or better persisting for at least 2 months, the dose interval was changed to once every 2 weeks (Q2W).
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 123 | 64
Completed | 0 | 0
Not Completed | 123 | 64
Not completed — Withdrawal by Subject | 7 | 7
Not completed — Death | 41 | 26
Not completed — Ongoing in the study | 75 | 31

BASELINE CHARACTERISTICS:
Population: Safety analysis set in each cohort included all enrolled participants in the respective cohort who received at least one dose of study intervention.
Groups:
- Cohort A: BCMA-naïve participants received subcutaneous elranatamab with a priming regimen of 12 milligrams (mg) on Cycle 1 Day 1 and 32 mg on Cycle 1 Day 4 followed by 76 mg weekly thereafter starting from Cycle 1 Day 8.
- Cohort B: BCMA-exposed participants received subcutaneous elranatamab with a priming regimen of 12 milligrams (mg) on Cycle 1 Day 1 and 32 mg on Cycle 1 Day 4 followed by 76 mg weekly thereafter starting from Cycle 1 Day 8.
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 123 | 64 | 187
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.1 (9.45) | 65.7 (9.42) | 66.6 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 34 | 89
  Male | 68 | 30 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 7 | 18
  Not Hispanic or Latino | 85 | 34 | 119
  Unknown or Not Reported | 27 | 23 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 1 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 2 | 11
  White | 72 | 44 | 116
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 26 | 17 | 43

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) by Blinded Independent Central Review (BICR) as Per International Myeloma Working Group (IMWG) Criteria
Description: ORR: % of participants with best overall response of confirmed stringent complete response (sCR), CR, very good partial response (VGPR) or PR per IMWG criteria. sCR: CR & normal serum free light chain (sFLC) ratio & absence of clonal cells in BMB/BMA by IH, IF, or flow cytometry. CR: negative immunofixation on serum & urine, disappearance of any soft tissue plasmacytoma & <5% plasma cells in BMA, if disease measurable by sFLC only, preceding criteria plus normal sFLC ratio. VGPR: Serum & urine M-protein detectable by immunofixation but not on electrophoresis; or >=90% reduction in serum M-protein & urine M-protein level <100mg/24h. PR: >=50% reduction in serum M-protein & reduction in 24h urinary M-protein by >=90% or <200 mg/24h. If serum & urine M-protein were unmeasurable, VGPR & PR: >=90% & >=50% decrease in difference respectively between involved & uninvolved sFLC levels & if present at baseline, >=90% & >=50% reduction in soft tissue plasmacytomas' size.
Time Frame: From date of first dose until confirmed disease progression, death, start of new anticancer therapy, whichever occurred first (up to approximately 16 months)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 123 | 64
Percentage of participants | 61.0 [51.8 to 69.6] | 34.4 [22.9 to 47.3]
Statistical Analysis 1: Comparison: Cohort A; Null hypothesis of ORR by BICR for cohort A was 30%; Test type: Other; p < 0.0001, Exact binominal
Statistical Analysis 2: Comparison: Cohort B; Null hypothesis of ORR by BICR for cohort B was 15%; Test type: Other; p < 0.0001, Exact binominal

2. Secondary Outcome: Cohort A Only: Objective Response Rate as Per IMWG Criteria by BICR for Participants With Extramedullary Disease (EMD) at Baseline
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Safety analysis set included all enrolled participants who received at least one dose of study intervention. Here, 'Overall Number of Participants Analyzed' signifies number of participants with EMD at baseline. This outcome measure was planned only in Cohort A.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 39
Percentage of participants | 38.5 [23.4 to 55.4]
Statistical Analysis 1: Comparison: Cohort A; Null hypothesis of ORR by BICR for cohort A was 12%; Test type: Other; p < 0.0001, Exact binominal

3. Secondary Outcome: Cohort A Only: Objective Response Rate as Per IMWG Criteria by BICR for Participants Without EMD at Baseline
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Safety analysis set included all enrolled participants who received at least one dose of study intervention. Here, 'Overall Number of Participants Analyzed' signifies number of participants without EMD at baseline. This outcome measure was planned only in Cohort A.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 84
Percentage of participants | 71.4 [60.5 to 80.8]
Statistical Analysis 1: Comparison: Cohort A; Null hypothesis of ORR by BICR for cohort A was 38%; Test type: Other; p < 0.0001, Exact binominal

4. Secondary Outcome: Duration of Response (DOR) as Per IMWG Criteria by BICR
Description: DOR: time from first documentation of objective response subsequently confirmed, until first documentation of confirmed PD or death due to any cause, whichever occurred first. PD= increase of >=25% from lowest value in >=1 of following (serum M-protein [absolute increase >=0.5g/dL]; serum M-protein increase >=1g/dL [when lowest M-protein >=5g/dL]; urine M-protein [absolute increase >=200mg/24h]; participants without measurable serum & urine M-protein levels, difference between involved & uninvolved sFLC levels [absolute increase >10mg/dL]; in participants without measurable serum, urine M-protein levels & involved sFLC levels: bone marrow plasma-cell % irrespective of baseline status [absolute increase >=10%]; appearance of new lesion,>=50% increase from nadir in SPD of >1 lesion, or >=50% increase in longest diameter of previous lesion >1cm in short axis; >=50% increase in circulating plasma cells [>=200cells/μL] if this is the only measure of disease.
Time Frame: From first documentation of objective response subsequently confirmed until confirmed PD or death due to any cause, or start of new anticancer therapy, whichever occurred first, or censoring (up to approximately 20.14 months)
Reporting Status: Not Posted, anticipated posting 2027-12

5. Secondary Outcome: Duration of Response as Per IMWG Criteria by Investigator Assessment
Description: as for outcome 4
Time Frame: as for outcome 4
Reporting Status: Not Posted, anticipated posting 2027-12

6. Secondary Outcome: Complete Response Rate (CRR) as Per IMWG Criteria by BICR
Description: CRR: % of participants with BOR of confirmed sCR/CR per IMWG criteria. sCR: CR & normal serum free light chain (sFLC) ratio & absence of clonal cells in BMB/BMA by IH, IF, or flow cytometry. CR: negative immunofixation on serum & urine, disappearance of any soft tissue plasmacytoma & <5% plasma cells in BMA, if disease measurable by sFLC only, preceding criteria plus normal sFLC ratio.
Time Frame: From date of first dose until confirmed disease progression, death, start of new anticancer therapy, whichever occurred first (up to approximately 20.14 months)
Reporting Status: Not Posted, anticipated posting 2027-12

7. Secondary Outcome: Complete Response Rate as Per IMWG Criteria by Investigator Assessment
Description: as for outcome 6
Time Frame: as for outcome 6
Reporting Status: Not Posted, anticipated posting 2027-12

8. Secondary Outcome: Objective Response Rate as Per IMWG Criteria by Investigator Assessment
Description: as for outcome 1
Time Frame: as for outcome 6
Reporting Status: Not Posted, anticipated posting 2027-12

9. Secondary Outcome: Duration of Complete Response (DOCR) as Per IMWG Criteria by BICR
Description: DOCR: time from first documentation of sCR/CR subsequently confirmed, until first documentation of confirmed PD or death due to any cause, whichever occurred first. PD= increase of >=25% from lowest value in >=1 of following (serum M-protein [absolute increase >=0.5g/dL]; serum M-protein increase >=1g/dL [when lowest M-protein >=5g/dL]; urine M-protein [absolute increase >=200mg/24h]; participants without measurable serum & urine M-protein levels, difference between involved & uninvolved sFLC levels [absolute increase >10mg/dL]; in participants without measurable serum, urine M-protein levels & involved sFLC levels: bone marrow plasma-cell % irrespective of baseline status [absolute increase >=10%]; appearance of new lesion,>=50% increase from nadir in SPD of >1 lesion, or >=50% increase in longest diameter of previous lesion >1cm in short axis; >=50% increase in circulating plasma cells [>=200cells/μL] if this is the only measure of disease.
Time Frame: From first documentation of sCR/CR subsequently confirmed until confirmed PD or death due to any cause, or start of new anticancer therapy, whichever occurred first, or censoring (up to approximately 20.14 months)
Reporting Status: Not Posted, anticipated posting 2027-12

10. Secondary Outcome: Duration of Complete Response (DOCR) as Per IMWG Criteria by Investigator Assessment
Description: as for outcome 9
Time Frame: From first documentation of objective sCR/CR subsequently confirmed until confirmed PD or death due to any cause, or start of new anticancer therapy, whichever occurred first, or censoring (up to approximately 20.14 months)
Reporting Status: Not Posted, anticipated posting 2027-12

11. Secondary Outcome: Progression Free Survival (PFS) as Per IMWG Criteria by BICR
Description: PFS was defined as the time from the date of first dose until confirmed PD or death due to any cause, whichever occurred first. PD= increase of >=25% from lowest value in >=1 of following (serum M-protein [absolute increase >=0.5g/dL]; serum M-protein increase >=1g/dL [when lowest M-protein >=5g/dL]; urine M-protein [absolute increase >=200mg/24h]; participants without measurable serum & urine M-protein levels, difference between involved & uninvolved sFLC levels [absolute increase >10mg/dL]; in participants without measurable serum, urine M-protein levels & involved sFLC levels: bone marrow plasma-cell % irrespective of baseline status [absolute increase >=10%]; appearance of new lesion,>=50% increase from nadir in SPD of >1 lesion, or >=50% increase in longest diameter of previous lesion >1cm in short axis; >=50% increase in circulating plasma cells [>=200cells/μL] if this is the only measure of disease.
Time Frame: From date of first dose until confirmed PD or death due to any cause, or start of new anticancer therapy, whichever occurred first, or censoring (up to approximately 20.14 months)
Reporting Status: Not Posted, anticipated posting 2027-12

12. Secondary Outcome: Progression Free Survival (PFS) as Per IMWG Criteria by Investigator Assessment
Description: as for outcome 11
Time Frame: as for outcome 11
Reporting Status: Not Posted, anticipated posting 2027-12

13. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time from the date of first dose until death due to any cause.
Time Frame: From the date of first dose until death due to any cause. Participants not known to have died were censored on the date of last known alive (up to approximately 20.14 months)
Reporting Status: Not Posted, anticipated posting 2027-12

14. Secondary Outcome: Time-to-Response (TTR) as Per IMWG Criteria by BICR
Description: TTR was defined, for participants with an objective response per IMWG criteria, as the time from the date of first dose to the first documentation of objective response that was subsequently confirmed.
Time Frame: as for outcome 1
Population: Safety analysis set in each cohort included all enrolled participants in the respective cohort who received at least one dose of study intervention. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 75 | 22
Months | 1.22 [0.89 to 7.36] | 1.92 [0.92 to 6.74]

15. Secondary Outcome: Time-to-Response (TTR) as Per IMWG Criteria by Investigator Assessment
Description: as for outcome 14
Time Frame: as for outcome 6
Reporting Status: Not Posted, anticipated posting 2027-12

16. Secondary Outcome: Minimal Residual Disease (MRD) Negativity Rate Per IMWG Sequencing Criteria
Description: MRD negativity rate was the percentage of participants with CR/sCR and with negative MRD per IMWG sequencing criteria.
Time Frame: as for outcome 6
Reporting Status: Not Posted, anticipated posting 2027-12

17. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) Graded by National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE was considered treatment-emergent relative to study intervention if the adverse event start date was during the on-treatment period (i.e. the time from the first dose of study intervention through the minimum of 90 days after last dose, or [start day of new anticancer therapy - 1 day]). CTCAE version 5.0 Grade 1: mild; Grade 2: moderate; Grade 3: severe or clinically significant; Grade 4: life-threatening; Grade 5: death.
Time Frame: From the date of first dose up to 90 days after last dose or new anticancer therapy whichever occurred first (up to approximately 20.14 months)
Reporting Status: Not Posted, anticipated posting 2027-12

18. Secondary Outcome: Number of Participants With Shift From Grade Less Than or Equal to (<=) 2 at Baseline to Grade 3 or 4 Post -Baseline in Laboratory Parameters by NCI CTCAE v 5.0
Description: CTCAE version 5.0 Grade 1: mild; Grade 2: moderate; Grade 3: severe or clinically significant; Grade 4: life-threatening.
Time Frame: as for outcome 17
Reporting Status: Not Posted, anticipated posting 2027-12

19. Secondary Outcome: Number of Participants With Cytokine Release Syndrome (CRS) Graded According to American Society for Transplantation and Cellular Therapy (ASTCT) Criteria
Description: CRS Grade 1: temperature >=38°C without hypotension or hypoxia; Grade 2: temperature >=38°C with hypotension not requiring vasopressors, and/or hypoxia requiring low-flow nasal cannula, facemask or blow-by; Grade 3: temperature >=38°C with hypotension requiring a vasopressor with or without vasopressin and/or hypoxia requiring high-flow nasal cannula, facemask, nonrebreather mask, or Venturi mask; Grade 4: temperature >=38°C with hypotension requiring multiple vasopressors (excluding vasopressin) and/or hypoxia requiring positive pressure (eg, continuous positive airway pressure [CPAP], bilevel positive airway pressure [BiPAP], intubation and mechanical ventilation); Grade 5: death.
Time Frame: as for outcome 17
Reporting Status: Not Posted, anticipated posting 2027-12

20. Secondary Outcome: Number of Participants With Immune Effector Cell-associated Neurotoxicity Syndrome (ICANS) Graded According to American Society for Transplantation and Cellular Therapy (ASTCT) Criteria
Description: ICANS Grade 1: immune effector cell encephalopathy (ICE) score 7-9, participant awakens spontaneously; Grade 2: ICE score 3-6, participant awakens to voice; Grade 3: ICE score 0-2, participant awakens only to tactile stimulus, any clinical seizure focal or generalized that resolved rapidly or nonconvulsive seizures on electroencephalography that resolve with intervention or focal/local edema on neuroimaging; Grade 4: ICE score 0 (participant is unarousable and unable to perform ICE), participant unarousable or requires vigorous or repetitive tactile stimuli to arouse, life-threatening prolonged seizure (>5 min), repetitive clinical or electrical seizures without return to baseline in between, deep focal motor weakness, diffuse cerebral edema on neuroimaging; decerebrate/decorticate posturing; cranial nerve VI palsy; papilledema, Cushing's triad; Grade 5: death. ICE: measures alterations in speech, orientation, handwriting, attention and receptive aphasia.
Time Frame: as for outcome 17
Reporting Status: Not Posted, anticipated posting 2027-12

21. Secondary Outcome: Serum Concentration of Elranatamab
Description: Total and free concentrations of Elranatamab on Cycle 4 Day 1 (C4D1) and Cycle 7 Day 1 (C7D1) were reported in this outcome measure.
Time Frame: Pre-dose on Day 1 of Cycle 4 and Pre-dose on Day 1 of Cycle 7
Population: The pharmacokinetic (PK) analysis set was a subset of safety analysis set and included participants who had at least one post dose concentration measurement. Here, "Overall Number of Participants Analyzed" signifies maximum participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 38 | 21
Nanograms per milliliter (ng/mL)
  Total elranatamab concentrations (C4D1): number analyzed (Participants) | 37 | 21
  Total elranatamab concentrations (C4D1) | 31100 (49) | 22840 (63)
  Total elranatamab concentrations (C7D1): number analyzed (Participants) | 29 | 9
  Total elranatamab concentrations (C7D1) | 37960 (47) | 29880 (77)
  Free elranatamab concentrations (C4D1) | 19090 (89) | 16170 (114)
  Free elranatamab concentrations (C7D1): number analyzed (Participants) | 29 | 9
  Free elranatamab concentrations (C7D1) | 32830 (81) | 29880 (49)

22. Secondary Outcome: Percentage of Participants With Positive Anti-Drug Antibody (ADA) and Neutralizing Antibodies (NAb) Against Elranatamab
Time Frame: From the date of first dose up to 20.14 months
Reporting Status: Not Posted, anticipated posting 2027-12

ADVERSE EVENTS:
Time Frame: From the date of first dose up to 90 days after last dose or start of new anticancer therapy whichever occurred first (up to approximately 20.14 months)
Description: Same event may appear as both non-SAE and SAE. What is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE. Safety analysis set evaluated. All-Cause Mortality:total number of deaths during study,from first dose of study drug and up to end of study are reported for all treated participants and included deaths which occurred after 90 days post last dose of study drug.
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 43/123 | 30/64
Serious Adverse Events (participants affected / at risk) | 84/123 | 44/64
Other Adverse Events (participants affected / at risk) | 123/123 | 63/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=123) | Cohort B (N=64)
Anemia (Blood and lymphatic system disorders) | 5 | 3
Aplasia pure red cell (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 0
Blindness (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Disease progression (General disorders) | 6 | 4
General physical health deterioration (General disorders) | 1 | 1
Inflammation (General disorders) | 1 | 1
Injection site reaction (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 1
Hepatitis fulminant (Hepatobiliary disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 16 | 7
Hypogammaglobulinaemia (Immune system disorders) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Adenovirus infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Aspergilloma (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 3 | 1
Bronchitis (Infections and infestations) | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 4
COVID-19 pneumonia (Infections and infestations) | 15 | 7
Cellulitis (Infections and infestations) | 0 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Cytomegalovirus infection reactivation (Infections and infestations) | 1 | 1
Device related bacteraemia (Infections and infestations) | 2 | 0
Device related sepsis (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1
Histoplasmosis (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 2 | 0
Lower respiratory tract infection viral (Infections and infestations) | 1 | 0
Parvovirus B19 infection (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 6 | 1
Pneumonia (Infections and infestations) | 9 | 3
Pneumonia adenoviral (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 3 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 1
Pneumonia influenzal (Infections and infestations) | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Post-acute COVID-19 syndrome (Infections and infestations) | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 2
Pyelonephritis acute (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 5 | 2
Septic shock (Infections and infestations) | 4 | 2
Sinusitis (Infections and infestations) | 3 | 0
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 2
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Parvovirus B19 test positive (Investigations) | 0 | 1
SARS-CoV-2 antibody test positive (Investigations) | 0 | 1
SARS-CoV-2 test positive (Investigations) | 2 | 2
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Sarcopenia (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Plasma cell myeloma refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 | 2
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 3 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 2
Renal failure (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypertension (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=123) | Cohort B (N=64)
Anaemia (Blood and lymphatic system disorders) | 58 | 39
Leukopenia (Blood and lymphatic system disorders) | 17 | 12
Lymphopenia (Blood and lymphatic system disorders) | 32 | 22
Neutropenia (Blood and lymphatic system disorders) | 59 | 24
Thrombocytopenia (Blood and lymphatic system disorders) | 36 | 27
Sinus tachycardia (Cardiac disorders) | 6 | 5
Tachycardia (Cardiac disorders) | 7 | 5
Abdominal pain (Gastrointestinal disorders) | 6 | 5
Constipation (Gastrointestinal disorders) | 16 | 11
Diarrhoea (Gastrointestinal disorders) | 47 | 18
Dry mouth (Gastrointestinal disorders) | 6 | 4
Nausea (Gastrointestinal disorders) | 32 | 9
Vomiting (Gastrointestinal disorders) | 19 | 8
Asthenia (General disorders) | 22 | 10
Chills (General disorders) | 10 | 2
Fatigue (General disorders) | 42 | 9
Injection site erythema (General disorders) | 9 | 5
Injection site reaction (General disorders) | 32 | 8
Oedema peripheral (General disorders) | 17 | 3
Pain (General disorders) | 5 | 5
Pyrexia (General disorders) | 27 | 11
Cytokine release syndrome (Immune system disorders) | 64 | 34
Hypogammaglobulinaemia (Immune system disorders) | 11 | 5
Pneumonia (Infections and infestations) | 7 | 6
Sinusitis (Infections and infestations) | 10 | 6
Upper respiratory tract infection (Infections and infestations) | 22 | 7
Urinary tract infection (Infections and infestations) | 8 | 6
Fall (Injury, poisoning and procedural complications) | 14 | 5
Alanine aminotransferase increased (Investigations) | 16 | 9
Aspartate aminotransferase increased (Investigations) | 18 | 7
Blood alkaline phosphatase increased (Investigations) | 8 | 2
Blood creatinine increased (Investigations) | 12 | 6
Blood lactate dehydrogenase increased (Investigations) | 7 | 4
SARS-CoV-2 test positive (Investigations) | 27 | 9
Weight decreased (Investigations) | 12 | 3
Decreased appetite (Metabolism and nutrition disorders) | 40 | 11
Hypercalcaemia (Metabolism and nutrition disorders) | 12 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 28 | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 11 | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 7 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 11
Dizziness (Nervous system disorders) | 13 | 2
Headache (Nervous system disorders) | 27 | 7
Insomnia (Psychiatric disorders) | 16 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 12 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 20 | 6
Erythema (Skin and subcutaneous tissue disorders) | 12 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 5
Rash (Skin and subcutaneous tissue disorders) | 10 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 6
Skin exfoliation (Skin and subcutaneous tissue disorders) | 13 | 6
Hypertension (Vascular disorders) | 10 | 3
Hypotension (Vascular disorders) | 12 | 5

LIMITATIONS AND CAVEATS:
Due to character limitation in outcome measure description, SPD definition is provided here. SPD was defined as the sum of the products of the maximal perpendicular diameters of measured lesions. Data for only those primary and secondary outcome measures whose analysis is complete and final have been reported. Data for remaining secondary outcome measures will be posted upon completion of analysis at secondary completion date.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/59/NCT04649359/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/59/NCT04649359/SAP_001.pdf